CLINICAL TRIAL: NCT01425489
Title: Biomarker for Krabbe Disease AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGI-CAL PROTOCOL
Brief Title: Biomarker for Krabbe Disease (BioKrabbe)
Acronym: BIOKRABBE
Status: Withdrawn | Type: Observational
Why Stopped: Transition into BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BK 06-2018
Record Dates: First submitted 2011-08-29; First posted 2011-08-30 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Krabbe Disease
Keywords: Krabbe Disease; Biomarker
MeSH Terms: conditions — Leukodystrophy, Globoid Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of mass-spectometry 10 ml EDTA blood and a dry blood spot filter card are taken. To proof the correct Krabbe diagnosis in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of Krabbe will be done as routine diagnostic.
  The analyses will be done at the Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Krabbe Disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Krabbe Disease from blood

DETAILED DESCRIPTION:
Krabbe disease is a rare, hereditary degenerative disorder of the central and peripheral nervous systems. It is characterized by the presence of globoid cells (cells that have more than one nucleus), the breakdown of the nerve's protective myelin coating, and destruction of brain cells. Krabbe disease is one of a group of genetic disorders called the leukodystrophies. These disorders impair the growth or development of the myelin sheath, the fatty covering that acts as an insulator around nerve fibers, and cause severe deterioration of mental and motor skills. Myelin is a complex substance made up of at least 10 different enzymes. Each of the leukodystrophies affects one (and only one) of these substances. Krabbe disease is caused by a deficiency of galactocerebrosidase, an essential enzyme for myelin metabolism. The disease most often affects infants, with on-set before age 6 months, but can occur in adolescence or adulthood.

Symptoms include irritability, unexplained fever, limb stiffness, seizures, feeding difficulties, vomiting, and slowing of mental and motor development. Other symptoms include muscle weakness, spasticity, deafness, and blindness.

Overall calculated European frequency is 1 case per 100,000 populations, with a higher reported incidence in Sweden of 1.9 cases per 100,000 populations. An unusually high incidence, 6 cases per 1000 live births, is reported in the Druze community in Israel.

New methods, like mass-spectrometry give a good chance to characterize in the blood (plasma) of affected patents specific metabolic alterations that allow to diagnose in the future the disease earlier, with a higher sensitivity and specificity. Therefore it is the goal of the study to develop new biochemical markers from the plasma of the affected patients helping to benefit the patient by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both gender from one year old
* The patient has a diagnosis of Krabbe Disease

EXCLUSION CRITERIA:

* No Informed consent from the patient or the parents before any study related procedures.
* Patients younger than one year
* The patient has no diagnosis of Krabbe Disease

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Krabbe Disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Krabbe disease from plasma | 24 month
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (5):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided